CLINICAL TRIAL: NCT03748277
Title: Prospective Comparative Study of Open and Minimally Invasive Surgical Techniques in the Treatment of Degenerative One-level Stenosis of Lumbar Spine
Brief Title: Comparison of Open and Minimally Invasive Surgical Techniques in the Treatment of Degenerative One-level Stenosis of Lumbar Spine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment terminated, all follow-up visits were canceled due to quarantine
Sponsor: Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15/11/18
Record Dates: First submitted 2018-11-15; First posted 2018-11-20 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-02

CONDITIONS: Spinal Stenosis Lumbar Canal With Neurogenic Claudication (Diagnosis)
Keywords: intraoperative procedures
MeSH Terms: conditions — Disease | interventions — Decompression

STUDY DESIGN:
Intervention Model Description: 1. group - decompression, MIS TLIF + Screw Fixation
  2. group - decompression, open fusion + Screw Fixation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive fusion (Experimental): Bilateral decompression using unilateral approach, MIS TLIF + screw fixation percutaneous
  Interventions: Procedure: Decompression; Procedure: MIS TLIF; Procedure: Screw Fixation
- Open Fusion (Active Comparator): Bilateral decompression, open fusion + screw fixation
  Interventions: Procedure: Decompression; Procedure: PLIF; Procedure: Screw Fixation

INTERVENTIONS:
Procedure: Decompression — Bilateral decompression
Procedure: PLIF — Traditional open surgery
  Arms: Open Fusion
Procedure: MIS TLIF — On the one side - Wiltse approach, on the other side - percutaneous
  Arms: Minimally invasive fusion
Procedure: Screw Fixation — Transpedicular Screw Fixation

SUMMARY:
The purpose of this study is to evaluate the clinical and radiological results of surgical treatment of one-level central stenosis of the lumbar spine using traditional open approach (PLIF) and a minimally invasive procedure (MIS TLIF). According to the hypothesis, we assume that unilateral approach of MIS TLIF allows for adequate bilateral decompression of one-level central stenosis of the lumbar spine. Using MIS TLIF it is possible to perform reliable fixation of a spine segment and the formation of a complete intervertebral bone fusion. The long-term clinical results of surgical treatment with minimally invasive technologies (MIS TLIF) and traditional open approach (PLIF) suspected to be comparable.

ELIGIBILITY:
Inclusion Criteria:

* syndrome of mono- or polyradicular compression of the nerve roots with / without a reflex pain syndromes, caused by stenosis of one lumbar spine segment;
* intermittent claudication caused by stenosis of one lumbar spine segment;
* one-level spine stenosis in combination with local segment instability or degenerative spondylolisthesis at the same spine segment, requiring fusion in only one lumbar segment

Exclusion Criteria:

* bilateral foraminal lumbar spine stenosis;
* lumbar spine stenosis more than one-level;
* spondylolisthesis II degree and more;
* sagittal imbalance;
* fusion the same lumbar spine segment after surgery previously;
* other diseases of the spine, including trauma, tumor and inflammatory diseases of the lumbar spine, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Day of hospital discharge (10-15 day after surgery)
  Oswestry Disability Index - patient-reported physical and household activity. Minimum - 0 (the worst result, patient is not physically active). Maximum - 50 (the best result).
  Improvement of ODI post-operatively as compared to baseline

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | 3, 6 and 12 months
  Oswestry Disability Index - patient-reported physical and household activity. Minimum - 0 (the worst result, patient is not physically active). Maximum - 50 (the best result).
  Improvement of ODI as compared to baseline
VAS (back, leg) | Day of hospital discharge (10-15 day after surgery), 3, 6 and 12 months
  Visual Analogue Scale (VAS) - patient-reported pain intensity (0 - no pain, 10 - unbearable pain).
  Improvement of VAS back- and leg pain intensity as compared to baseline
Surgery duration | Day of surgery
  Surgery duration, in minutes
Blood loss | Day of surgery
  Blood loss, in milliliter
MRI capacity spine canal | Day of hospital discharge (10-15 day after surgery)
  Changes of spine canal capacity of spine segment, in sq. cm., as compared to baseline
Bone fusion | 12 months
  Intervertebral bone fusion formation, in degree (I, II, III or IV degree according to Tan)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr V Krutko, PhD, MD, Principal Investigator — Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan, Neurosurgery Department
Locations (1):
- Novosibirsk Research Institute of Traumatology and Orthopaedics n.a. Ya.L. Tsivyan, Novosibirsk, Russia